CLINICAL TRIAL: NCT01956214
Title: Efficacy of Functional Electrical Stimulation Exercise Training in Hemodialysis Patients
Brief Title: Functional Electrical Stimulation (FES) Exercise Training in Hemodialysis Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB#: 12309
Record Dates: First submitted 2013-04-17; First posted 2013-10-08 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2014-08

CONDITIONS: Complication of Dialysis
Keywords: hemodialysis; exercise; electrical stimulation
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FES exercise (Experimental): Participants will receive FES
  Interventions: Other: FES Exercise
- Mock FES exercise (Sham Comparator): participant will receive Mock FES
  Interventions: Other: Mock FES Exercise

INTERVENTIONS:
Other: FES Exercise — receive FES while exercising
  Arms: FES exercise
Other: Mock FES Exercise — participants will receive Mock FES
  Arms: Mock FES exercise

SUMMARY:
Both strength training and endurance exercise training are commonly prescribed to improve strength and function in patients with physical limitations caused by chronic disease or disability including chronic kidney disease (CKD). Individuals with CKD often have low physical function due to progressive declines in the performance of their kidneys. The low physical function leads to physical inactivity, which exacerbates these functional declines and promotes cardiovascular disease and bone disorders. In addition, severe functional limitations in some patients prevent them from exercising at a great enough intensity to provide significant benefits. As a result, alternative strategies are needed to maximize the benefits of exercise while decreasing injury risk.

DETAILED DESCRIPTION:
Both strength training and endurance exercise training are commonly prescribed to improve strength and function in patients with physical limitations caused by chronic disease or disability including chronic kidney disease (CKD). Individuals with CKD often have low physical function due to progressive declines in the performance of their kidneys. The low physical function leads to physical inactivity, which exacerbates these functional declines and promotes cardiovascular disease and bone disorders. In addition, severe functional limitations in some patients prevent them from exercising at a great enough intensity to provide significant benefits. As a result, alternative strategies are needed to maximize the benefits of exercise while decreasing injury risk.

A new form of exercise, functional electrical stimulation (FES)-enhanced cycling has been shown to increase muscle size and strength in patients with severe disabilities, particularly spinal cord injury (SCI). It is based on the application of electrical stimulation to the nerves that innervate the paralyzed weak muscles in order to generate muscle contraction. FES has been used to stimulate leg muscles to pedal a cycle or to enable partial weight-supported walking as an activity based rehabilitation therapy. FES cycling involves exercising using a motor-assisted cycle coupled with electrical stimulation to up to five muscles in the leg. There are well-documented benefits of FES-induced exercise in SCI patients including clinically significant increases in muscle mass, blood flow, bone density, and bowel and bladder function. A few pilot studies have also demonstrated that FES therapy has the potential to improve function in other disabled populations, including chronic heart failure and stroke patients. However, its effects in other populations with significant physical impairments, including CKD patients, have yet to be established.

The objective of the proposed research is to evaluate the effects of FES-cycling training on measures related to physical function, quality of life (QOL), heart disease, and bone health in patients with renal failure receiving dialysis therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 31-85 years
2. Must receive hemodialysis treatment at least 3 days per week
3. Must be willing to be randomized to the control or FES-cycle groups
4. Must receive medical clearance from a Nephrologist at their dialysis clinic to participate
5. Must have evidence of impaired mobility on the FES Screening Form, attached. The FES Screening Form inclusion criterion consist of a questionnaire of five tasks with a relative difficulty scale for the completion of each task. Participants will be included in the study if they indicate "some" or more difficulty at any task on the questionnaire.

Exclusion Criteria:

1. On dialysis treatment for less than 3 months.
2. Body weight of greater than 400 pounds. (weight limitations on the DXA table)
3. Unstable angina, recent (less than 3 months) myocardial infarction or stroke (these conditions may not enable the patient to tolerate the proposed exercise training).
4. Implanted electronic pacing or defibrillation device, vagus nerve stimulator, or unstable vital signs.(the safety of electrical stimulation under these conditions is not known).
5. Metal implants underneath or near the muscle groups which are to be stimulated.
6. Pregnancy (the safety of stimulation during pregnancy is not known) - a section on the ICD has been created for women to initial to indicate they are NOT pregnant or planning on becoming pregnant over the course of the study.
7. Lower limb amputation.

On the PAR-Q form, if the participant answers YES to the question: "Has your doctor ever said that you have a heart condition and that you should only do physical activity recommended by a doctor?", they will be excluded from the study.

We will also use answers on the Medical History Form to help us evaluate the exclusion criteria. Answers to the following questions will either be exclusionary, or require further follow-up with a physician prior to being allowed to participate:

Question 1: "Do you ever get chest pains while at rest and/or during exertion?", and Question 4: "…was your heart attack within the last year?" An answer of YES to either question will require that the individual obtain a comprehensive physical exam by their physician prior to being allowed to participate.

Question 10: Has your physician ever specifically told you not to do "heavy" or "hard" exercise? An answer of YES will require a physical exam.

Under "Medical History" (top of page 2 of Medical History Form), or "Present Symptoms Review" (top of page 3) a check by "chest pain or pressure" will require a physical exam.

Under "Present Symptoms Review (top of page 3), a check by any of the following will lead to exclusion: Implanted electronic pacing or defibrillation device; vagus nerve stimulator; metal implants in the legs; or unstable vital signs.

Ages: 31 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-12; Primary Completion 2015-12 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
physical function | Three months
  muscle strength, functional fitness testing, shuttle walk test, balance and gait kinematics

OTHER OUTCOMES:
quality of life (QOL) | three months
  questinnaire
heart disease | three months
  arterial and cardiac measures
bone health | three months
  DXA scan for bone mineral density, body composition, vascular calcification

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Wilund, PhD, Principal Investigator — UIUC
Locations (1):
- Champaign Urbana Dialysis Center, Urbana, Illinois, United States